CLINICAL TRIAL: NCT04881110
Title: Effects of the Glucagon Like-peptide 1 (GLP-1) Receptor Agonist Liraglutide on Lower Limb Perfusion in People With Type 2 Diabetes and Peripheral Artery Disease: a Randomized Controlled Trial
Brief Title: Liraglutide and Peripheral Artery Disease
Acronym: STARDUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Katherine Esposito, Professor of Endocrinology and Metabolic Diseases, Head of Unit of Diabetes, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2_0401_2021
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Peripheral Arterial Disease
Keywords: Type 2 diabetes; Liraglutide; Transcutaneous Oxygen Tension; Peripheral arterial disease; Inflammation; Angiogenesis; Endothelial Dysfunction; Diabetic microvascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Arterial Disease; Inflammation | interventions — Liraglutide; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide group (Experimental): Patients in this arm will receive liraglutide, according to the current clinical practice.
  Interventions: Drug: Liraglutide
- Control group (Other): Patients in this arm will be strictly monitored with optimization of the therapy for atherosclerosis major risk factors.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Liraglutide — Patients in this arm will receive one daily subcutaneous injection of liraglutide. The starting dose is 0.6 mg/dl per day. The dose has to be increased to 1.2 mg/dl per day after the first week of treatment and to 1.8 mg/dl after the second one.
  Other Names: Intervention group
  Arms: Liraglutide group
Other: Control — Patients in this arm will be strictly monitored for atherosclerosis major risk factors, such as hypertension and dyslipidemia, and treated according to current clinical practice.
  Other Names: Control group
  Arms: Control group

SUMMARY:
STARDUST is an open-label, two-arm randomized controlled trial, aimed at evaluating the effects of liraglutide on peripheral perfusion, as compared with the aggressive treatment of cardio-metabolic risk factors, in people with type 2 diabetes and peripheral artery disease. The potential benefits for participants in the study include the possibility of improving peripheral perfusion with drugs that have been evaluated as effective in controlling diabetes and safe and protective for cardiovascular health.

The primary outcome of the study is the change of peripheral transcutaneous oxygen tension between groups at three and six months. Participants in the study will be followed for 6 months in order to evaluate the effects of liraglutide and the change of other secondary outcomes.

DETAILED DESCRIPTION:
An 18-month extension of the follow-up will be performed for all the study population, according to guidelines and good clinical practice. The follow-up will include the glyco-metabolic parameters and the main cardiovascular risk factors, including TcPO2 assessment.

Data from this extended observation will be collected for additional analyses (mostly regarding the durability of the effects). Individuals who will be lost during follow-up and/or discontinue or modify the glucose-lowering treatment will be excluded from the analyses.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes within at least 6 months
* peripheral arterial disease documented within al least 1 year by doppler ultrasound, angio-CT or arteriography
* peripheral transcutaneous oxygen pressure between 30 and 49 mmHg on anterior and/or posterior tibial arteries
* Hba1c 6,5-8%
* treatment of diabetes with metformin, insulin and/or sulfonylurea

Exclusion Criteria:

* diagnosis of type 1 diabetes
* current treatment with GLP-1 receptor agonists (GLP-1RAs) or dipeptidyl peptidase -4 (DPP-4) inhibitors
* GLP-1RAs allergy or intolerance
* participation to other clinical studies
* history of pancreatitis, thyroid disease, diabetic gastroparesis or inflammatory bowel disease
* current or planned pregnancy
* acute myocardial infarction and/or acute cerebrovascular disease within 14 days from the screening visit
* planned revascularization procedure
* renal function with estimated glomerular filtration rate (eGFR) below 15 ml/min
* history of cancer and/or oncological treatment within 5 years from the screening visit
* current treatment with corticosteroids
* psychiatric or other clinical conditions which may interfere with the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Esposito, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Unit of Endocrinology and Metabolic Diseases and Unit of Diabetes, University of Campania Luigi Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caruso P, Maiorino MI, Bellastella G, Esposito K, Giugliano D. Pleiotropic effects of GLP-1 receptor agonists on peripheral artery disease: Is there any hope? Diabetes Metab Res Rev. 2023 Oct;39(7):e3627. doi: 10.1002/dmrr.3627. Epub 2023 Mar 4. No abstract available. PMID 36812501
- [Derived] Caruso P, Maiorino MI, Longo M, Porcellini C, Matrone R, Digitale Selvaggio L, Gicchino M, Carbone C, Scappaticcio L, Bellastella G, Giugliano D, Esposito K. Liraglutide for Lower Limb Perfusion in People With Type 2 Diabetes and Peripheral Artery Disease: The STARDUST Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e241545. doi: 10.1001/jamanetworkopen.2024.1545. PMID 38470420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide Group | Control Group
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide Group | Control Group | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [62.5 to 72.0] | 65.0 [60.0 to 73.0] | 65 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 11.0 [5.5 to 25] | 10.0 [3 to 30] | 10 [4 to 30]
TcPO2 [Mean (Standard Deviation); unit: mmHg] | 40.0 (5.9) | 40.5 (5.7) | 40.3 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Transcutaneous Oxygen Pressure
Description: Transcutaneous oxygen pressure (mmHg) on the lowest value recorded on anterior or posterior tibial artery after 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mmHg | 54.2 (5.9) | 43.4 (4.8)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [8.0 to 14.5]; To evaluate the change of variables over time, we subtracted the values at the start from values at the end. A 2-sample t test was used to compare differences between the interventions. The χ2 test was used for comparing proportions of participants in the 2 groups who reached the primary end point after the intervention. Relative risks (RRs) and 95%Cis were calculated to demonstrate the relationship between the intervention and the achievement of the primary end point. A 2-sided P < .05 was considered statistically significant
Statistical Analysis 2: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p < 0.001, Chi-squared; Risk Ratio (RR) = 1.91, 95% CI 2-sided [1.26 to 2.90]; [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: HbA1c Glucose Control
Description: HbA1c values after 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
percentage of HbA1c | 6.7 (0.7) | 6.8 (0.8)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to 0.01]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Glucose Control
Description: fasting glucose differences between groups
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mg/dL | 118.5 [91 to 132.5] | 117 [98 to 122]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.52, t-test, 2 sided; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-14.3 to 7.4]; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Weight Change
Description: Weight value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
Kg | 78.5 (14.4) | 80.7 (12.5)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.33, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.6 to 1.2]; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: BMI Change
Description: BMI value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
Kg/m2 | 28.7 (4) | 27.7 (4.4)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.1]; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Waist Circumference Change
Description: Waist circumference value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
cm | 108.9 (10.3) | 104.1 (11.6)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.81, t-test, 2 sided; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-2.8 to 3.5]; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Systolic Blood Pressure Change
Description: systolic blood pressure value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mmHg | 130 [120 to 130] | 130 [125 to 140]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.99, t-test, 2 sided; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-5.8 to 5.8]; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: Lipid Profile
Description: total cholesterol after 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mg/dL | 142.3 (40.6) | 158.8 (55.1)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-32.6 to 22.9]; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: C-reactive Protein (CRP) Change
Description: CRP value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mg/dL | 0.5 (0.5) | 0.8 (0.5)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.07]; [other analysis details as in outcome 1, analysis 1]

10. Secondary Outcome: Renal Function
Description: creatinine levels after 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mg/dL | 1 [0.8 to 1.2] | 0.8 [0.8 to 1]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.12, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.04 to 0.3]; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: Estimated Glomerular Filtration Rate
Description: estimated glomerular filtration rate after 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
mL/min/1.73 m^2 | 71 (18.4) | 74.7 (13.4)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-8.5 to 2.3]; [other analysis details as in outcome 1, analysis 1]

12. Secondary Outcome: Angiogenesis
Description: vascular endothelial growth factor (VEGF) after 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
pg/mL | 124 [77.5 to 188] | 68.4 [52.2 to 80.8]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 87.4, 95% CI 2-sided [59.9 to 115.1]; [other analysis details as in outcome 1, analysis 1]

13. Secondary Outcome: Ankle-brachial Index (ABI) Change
Description: ABI value after 6 months minus value at baseline ABI evaluation was obtained dividing the leg systolic pressure by the arm systolic pressure, both detected through a doppler probe and a sphygmomanometer.
  Normal ABI ranges from 1.0 to 1.4. ABI values above 1.4 suggest a noncompressible calcified vessel. ABI value below 0.9 is considered diagnostic of PAD.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
ratio | 0.9 [0.9 to 1] | 1 [0.9 to 1.1]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.09 to 0.01]; [other analysis details as in outcome 1, analysis 1]

14. Secondary Outcome: Sexual Hormonal Profile
Description: Sexual hormone binding protein after 6 months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
nmol/L | 45 [34.1 to 51.7] | 49.5 [44.5 to 66.2]
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [-0.6 to 18.1]; [other analysis details as in outcome 1, analysis 1]

15. Secondary Outcome: Male Sexual Function
Description: Erectile function (IIEF-5) score at 6 months Male patients will perform a self-assessment test (IIEF-5) of their erectile function and overall satisfaction with sexual life, referring to the previous 6 months.
  Erectile dysfunction (ED) will be classified based on the total questionnaire score. The highest score available is 25, the lowest is 0. Any score ranging from 25 and 22 refers to the absence of ED.
  Any score ≤ 21 will indicate the presence of ED [mild (score 21-17), mild-moderate (score 16 -12), moderate (score 11-8) and severe (score 7-1)].
  The IIEF-5 questionnaire will be administered at visit 2 (week 0) and at the end of the study (week 24).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 21 | 22
score on a scale | 12.4 (5.7) | 12.5 (4.6)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.09 to 2.6]; [other analysis details as in outcome 1, analysis 1]

16. Secondary Outcome: Female Sexual Function
Description: Female sexual function (FSFI) after 6 months Female sexual function will be studied through the FSFI questionnaire which assesses sexual activity over the past 4 weeks and includes 19 questions. The questionnaire will investigate six distinct domains (sexual desire, arousal, lubrication, orgasm, satisfaction and pain), and provide a total score indicative of global sexual function.
  Points are assigned for each answer (from 1 to 5 for 1-2 questions, from 0 to 5 for 3-19): the sum of the scores for each domain is multiplied by a domain factor (desire 0.6, arousal 0.3, lubrication 0.3 orgasm 0.4, satisfaction 0.4, pain 0.4). The six domain scores are added up, and the total score may vary from 2.0 to 36.0 points.
  A total FSFI score < 26.55 will be used to classify the presence of female sexual dysfunction. The FSFI questionnaire will be administered at visit 2 (week 0) and at the end of the study (week 24).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 6 | 6
score on a scale | 20.4 (1.4) | 21.2 (1.3)

17. Secondary Outcome: 6-minute Walking Test
Description: 6-minutes walking distance after 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Liraglutide Group | Control Group
Number analyzed (Participants) | 27 | 28
meters | 364 (13.7) | 340 (11.5)
Statistical Analysis 1: Comparison: Liraglutide Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 25.1, 95% CI 2-sided [21.8 to 28.3]; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events occurred.
Arm/Group | Liraglutide Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT04881110/Prot_000.pdf